CLINICAL TRIAL: NCT01511120
Title: Ringer's Acetat Versus Balanced Hydroxyethyl-starch as Primesolution in the Heart-lung Maschine During Cardio-pulmonary-bypass. Postoperatively Fluid Balance and Cardiac Function
Brief Title: The Effect on Fluid Balance After Cardiac Surgery After Use of Two Different Priming Protocols
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011/498
Record Dates: First submitted 2011-12-07; First posted 2012-01-18 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tetraspan (Active Comparator)
  Interventions: Drug: Tetraspan; Drug: acetated Ringer's solution

INTERVENTIONS:
Drug: Tetraspan
  Other Names: Tetraspan® (HES 130/0,42 , 6%),; B. Braun Medical AS; Kjernåsveien 13 B; 3142 Vestskogen
Drug: acetated Ringer's solution

SUMMARY:
"The impact on fluid loading after cardiac surgery by use of two different priming solution"

Fluid overloading with oedema formation is a regular finding following on-pump cardiac surgery and may contribute to postoperative organ dysfunction. Myocardial oedema has been reported to impair both systolic and diastolic function. An association between intraoperative fluid loading and postoperative adverse outcome has been demonstrated in cardiac patients.

The investigators have experience with the use of both colloides and combination fluids (hypertonic saline/colloides) in several experimental studies (pigs). In one animal study the investigators used colloides as an additive to the CPB-prime. The investigators observed reduced fluid leakage and less total tissue water in several organs.

The planned study includes patients scheduled for coronary artery bypass, and who have no co-morbidity. The patients will be randomized to receive either Tetraspan® (HES) or acetated Ringer's solution in the CPB-prime. Accurate accounts of fluid additions, blood loss and diuresis will be kept. Determination of cardiac output (C.O.), intrathoracic blood volume (ITBV), extravascular lung water (EVLW) and global end diastolic volume (GEDV) will be monitored by use of the transpulmonary thermodilution technique PiCCO®plus system.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CABG,
* EF(ejection fraction) more than 40%

Exclusion Criteria:

* Reduced EF (less than 40%) EVF less than 30%,
* Estimated GFR less than 60%,
* BMI less than 18 or more than 32

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Reduction of organ edema and improved organ function | 6-hours postoperatively
  As a target of effect the investigators have chosen to study improvements for organ function.Indexed values for cardiac output(CI) measured by the PICCO system will be a parameter for heart function, andf lung function will be measured by EVLWI(extravascular lungwater index).paO2/FiO2-ratio and time spent in respirator.Additionally a strict account for fluid balance will be kept.

CONTACTS AND LOCATIONS:
Locations (1):
- Hjerteavdelingen, thoraxkirurgisk seksjon, Haukeland Universitetssykehus, Bergen, Norway

REFERENCES:
- [Derived] Svendsen OS, Farstad M, Mongstad A, Haaverstad R, Husby P, Kvalheim VL. Is the use of hydroxyethyl starch as priming solution during cardiac surgery advisable? A randomized, single-center trial. Perfusion. 2018 Sep;33(6):483-489. doi: 10.1177/0267659117746235. Epub 2017 Dec 4. PMID 29199540